CLINICAL TRIAL: NCT02458976
Title: Pulsed-dye Laser Treatment Prior to Surgical Excision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Professor of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015P000196
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Cicatrix
Keywords: Scar; Pulsed-dye laser; PDL
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDL (Experimental): Pre-treatment of surgical area with PDL
  Interventions: Device: PDL

INTERVENTIONS:
Device: PDL

SUMMARY:
This prospective pilot study will investigate whether use of a pulsed dye laser (PDL) prior to surgical excision can improve the appearance and symptoms of scars. The primary outcome measurement for the study is the quality of the scar in areas pre-treated with PDL vs. control (cryogen spray only). For this study, subjects who are scheduled for a dermatologic surgical excision will have half of the surgical area pre-treated with PDL and the other half pre-treated with cryogen spray.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ages between 18 and 65 years, who are scheduled for a dermatologic surgical excision
* Subjects requiring surgical excisions for any condition
* Subjects with any Fitzpatrick skin type
* Willingness to participate in the study
* Willingness to receive experimental treatment
* Informed consent agreement signed by the subject
* Willingness to follow the follow-up schedule
* Willingness to not use any other scar treatments during the study period (i.e scar massage, over-the-counter silicone pads, intralesional steroid of 5-fluorouracil injections, laser treatments)

Exclusion Criteria:

* Pregnancy
* Prior scar in area to be treated
* Known photoallergy to visible light (i.e polymorphous light eruption)
* Subject is unable to comply with treatment or follow-up visits
* Subject with a history of being on photosensitive medications for the past 3 months (thiazides [used to treat high blood pressure], tetracyclines, fluoroquinolones griseofulvin or sulfonamides [used to treat infections], sulfonylureas [used to treat diabetes], calcium channel blockers [used to treat hypertension], phenothiazines [used to treat serious emotional problems]).
* Known autoimmune disease (some autoimmune diseases can lead to sensitivity to light, such as lupus erythematosus)
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Scar appearance | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: R R Anderson, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No